CLINICAL TRIAL: NCT01478074
Title: A Single-center Open-label Phase I Study of ALT-801 for ex Vivo Maturation and in Vivo Retargeting of Haploidentical Natural Killer Cells Delivered Following Fludarabine, Cytarabine, and G-CSF in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: ALT-801-activated Natural Killer Cells After FLAG Induction for Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The treatment planned was determined to be of low feasibility as no subject was found eligible and able to enroll after screening over 30 subjects
Sponsor: Altor BioScience (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-02-08
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed leukemia; Refractory leukemia; Natural Killer Cells; Adoptive immunotherapy; NK cell infusion; Haploidentical; KIR mismatch; Fludarabine; Cytarabine; Ara-C; ALT-801
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Granulocyte Colony-Stimulating Factor; Cytarabine; fludarabine; Cell Count; ALT-801

ARMS (1):
- FLAG + NK Cells + ALT-801 (Experimental)
  Interventions: Drug: G-CSF; Drug: Cytarabine; Drug: Fludarabine; Biological: Donor Natural Killer (NK) cells; Biological: ALT-801

INTERVENTIONS:
Drug: G-CSF — 5 mcg/kg daily from day -7 until post-nadir ANC > 1000
Drug: Cytarabine — 2 g/m2 daily from day -6 through -2
Drug: Fludarabine — 30 mg/m2 daily from day -6 through -2
Biological: Donor Natural Killer (NK) cells — Infused once on day 0. Four cohorts of escalating doses receiving 0, 1, 10, or 20 x 10^6 cells/Kg
Biological: ALT-801 — 0.04 mg/kg IV thrice weekly for 8 doses beginning day +2

SUMMARY:
This is a single-center open-label phase I clinical trial of delivering haploidentical natural killer (NK) cells matured ex vivo with ALT-801 followed by intravenous infusions of ALT-801 in patients with relapsed/refractory Acute Myeloid Leukemia (AML). The study will be conducted at M.D. Anderson Cancer Center (MDACC) and MDACC Children's Cancer Hospital in Houston, Texas.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (SCT) is an effective treatment for acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). For patients transplanted in first remission or with low risk MDS, approximately 60% of patients have achieved long-term disease free survival. Patients with relapsed leukemia have a poorer outcome; the long-term disease free survival rate for relapsed AML is 5-10% without hematopoietic stem cell transplantation (HSCT). With HSCT, survival after relapse approaches 40%, but success depends greatly on whether patients are in remission at the time of transplant. Many relapsed patients have refractory chemoresistant disease and never attain remission to be eligible for potentially curative HSCT, or develop significant complicating comorbidities during the prolonged intensive reinduction of their disease. Thus, improved strategies for achieving remission in relapsed patients prior to transplantation are critical to improving the survival of these patients. Relapsed/refractory AML requires remission prior to allogeneic HSCT for optimal survival, but responds poorly to chemotherapy. Human leukocyte antigen (HLA)-haploidentical, NK-enriched peripheral blood cell infusions may augment induction chemotherapy in patients with poor prognosis AML, but there are significant toxicities related to the IL-2 infusions given for optimal NK cell activity. The purpose of this trial is to estimate the toxicity and feasibility of treating relapsed/refractory AML with FLAG chemotherapy followed by haploidentical donor-derived natural killer (NK) cells using ALT-801 for ex vivo and in vivo NK cell activation as an alternative to interleukin-2 (IL-2).

ALT-801 is a genetically engineered fusion protein, that is, a single protein made by combining the DNA of two or more different genes. ALT-801 is a combination of IL-2 (an important protein for stimulating immune cells) and a binding portion that recognizes tumor cells.

The primary objective of this study is to evaluate the safety and feasibility of an infused allogeneic donor NK cell product and ALT-801 following a FLAG preparative regimen to treat relapsed/refractory acute myelogenous leukemia. The primary endpoint for toxicity is the absence of NK cell Product or ALT-801-related grade 2 toxicity, excluding grade 2 fever, rigor/chills, fatigue, vomiting/nausea, pruritus/itching, electrolyte imbalance, hypoalbuminemia or lymphopenia within 21 days of the ALT-801 or NK cell product infusion. The primary endpoint of feasibility is defined as being able to infuse NK-cells at the maximum tolerated cell dose or the highest dose level on day 0 and complete all 8 planned doses of ALT-801, with a safety that does not exceed toxicity limits, in greater than or equal to 7 of 10 subjects.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Patients with relapsed AML, including those with CNS disease or previous hematopoietic stem cell transplantation, or primary refractory AML (primary AML that has failed remission to at least two cycles of induction therapy)
2. For patients of Cohorts 2 to 4, availability of a haploidentical family peripheral blood stem cell donor selected for best possible KIR reactivity
3. Patient is between 2 and 59 years of age, inclusive
4. Patient must have recovered from the treatment-related toxicities of prior cytotoxic agents received in the 4 weeks prior to beginning treatment on this protocol, with the exception of cytopenias resulting from persistent disease, and alopecia
5. Zubrod performance scale (Refer to Appendix C) ≤ 2 or Lansky (Refer to Appendix D) > 60
6. Adequate renal function defined as:

   * For adults serum creatinine < 2 mg/dL
   * For children serum creatinine < 2 mg/dL or < 2 times upper limit of normal (ULN) for age (which ever is less) If abnormal creatinine level, 24h creatinine clearance > 60 mL/min/1.73m^2
7. Adequate liver function, defined as: Total bilirubin ≤ 2 mg/dL and SGPT (ALT) ≤ 2.5 x ULN for age (unless Gilbert's disease or abnormal liver function due to primary disease)
8. Pulmonary symptoms controlled by medication and pulse oximetry> 92% room air
9. New York Heart Association classification < III
10. Negative serum test to rule out pregnancy within 2 weeks prior to registration in females of childbearing potential (non childbearing potential defined as premenarchal, greater than one year post-menopausal, or surgically sterilized)
11. Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator
12. Negative serology for human immunodeficiency virus (HIV)

Recipient Exclusion Criteria:

1. Investigational therapies in the 4 weeks prior to beginning treatment on this protocol
2. Congestive heart failure < 6 months prior to screening
3. Unstable angina pectoris < 6 months prior to screening
4. Myocardial infarction < 6 months prior to screening

Donor Inclusion Criteria:

1. Related to recipient (sibling, parent, offspring, offspring of a sibling)
2. HLA-haploidentical to recipient (need not be re-tested if already performed previously, provided copies of the original results are available)
3. Able and willing to undergo apheresis
4. Willing to donate blood for baseline chimerism assessment
5. Negative serum test to rule out pregnancy within two weeks prior to registration in females of childbearing potential (non childbearing potential defined as premenarchal, greater than one year post-menopausal, or surgically sterilized)
6. Donor must meet institutional eligibility criteria for allogeneic blood stem cell donation including infectious disease screening panel (Hepatitis B, Hepatitis C, HIV, CMV, and West Nile Virus) and CBC, differential and platelet studies
7. Donor must meet stem cell donor eligibility criteria as set forth in 21 CFR 1271 subpart C
8. The preferred Donor will be selected as the most alloreactive of the available haploidentical related donors on the basis of predicted NK cell alloreactivity using Recipient and Donor HLA type. If necessary, the best of equally alloreactive donors will be determined by Donor KIR type. NK alloreactivity is defined as o A KIR gene is present on the Donor NK cells for which

   * the HLA haplotype (KIR ligand) for the KIR receptor in question is absent in the Recipient, and
   * the HLA haplotype (KIR ligand) for the KIR receptor in question is present in the Donor

Donor Exclusion Criteria:

1. Active infection (defined as on antimicrobial therapy and/or febrile)
2. Pregnant females
3. Breast-feeding females

Ages: 2 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of NK cells | 18 months
  Determined by the maximum tolerated dose of NK cells that can be given in combination with ALT-801 with less than 1/3 of patients experience dose-limiting toxicities related to the NK cells or ALT-801.
Safety of delivering NK cells and ALT-801 in combination with FLAG | 6 months after study completes accrual
  Determined by whether the maximum tolerated dose of NK cells can be given in combination with ALT-801 and FLAG chemotherapy without exceeding a rate of 0.28 for >= Grade 3 toxicities (10% above that of FLAG therapy alone) during the treatment period.

SECONDARY OUTCOMES:
Activation status of NK cells following activation with ALT-801 | 6 months after study completes accrual
  Activation status of ALT-801-activated NK cells will be determined by measuring NK cell degranulation against standardized targets and comparing with freshly-obtained NK cells.
In vivo persistence and function of haploidentical NK cells activated with ALT-801. | 6 months after study completes accrual
  Determined by measuring levels of donor NK cells in the blood and their degranulation against standardized targets.
Overall response to this regimen | 6 months after study completes accrual
  Determined according to AML Response Criteria in NCCN Practice Guidelines for Oncology v.1.2008.
Rate of stem cell transplantation and the time-to-transplantation | 6 months after study completes accrual
  Determined by reporting how often and at what time patients achieve sufficient remission and health status to receive hematopoietic stem cell transplantation as definitive therapy after receiving this combination of chemotherapy, cellular therapy, and immune therapy.
ALT-801 immunogenicity | 6 months after study completes accrual
  Determined by measuring levels of anti-ALT-801 antibodies in serum before treatment and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hing C Wong, PhD, Study Director — Altor BioScience
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States